CLINICAL TRIAL: NCT02289885
Title: Knowledge, Attitude and Practice About Focused Assessment With Sonography in Trauma Among Paramedics. Randomized Crossover Manikin Trial
Brief Title: FAST Examination During Emergency Practice
Acronym: FAST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FAST/2014/02
Record Dates: First submitted 2014-11-07; First posted 2014-11-13 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Trauma; Ultrasonography
Keywords: trauma; examination; knowledge; paramedic
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- normal model patient (Experimental): Images of the ultrasound window were captured to disk and later evaluated by an expert in emergency medicine. In this study, the FAST examination was measured to the perihepatic space (also called Morison's pouch or the hepatorenal recess), perisplenic space, pericardium, and the pelvis.
  Interventions: Device: SonoScape
- ascites positive model patient (Experimental): Images of the ultrasound window were captured to disk and later evaluated by an expert in emergency medicine. In this study, the FAST examination was measured to the perihepatic space (also called Morison's pouch or the hepatorenal recess), perisplenic space, pericardium, and the pelvis.
  Interventions: Device: SonoScape

INTERVENTIONS:
Device: SonoScape — Ultrasonography device
  Other Names: SonoScape S6 Portable Ultrasound Machine

SUMMARY:
The study evaluates the knowledge, attitude and practice about Focused Assessment with Sonography in Trauma among emergency medicine practitioners in Poland.

ELIGIBILITY:
Inclusion Criteria:

* Paramedics currently practicing in a Polish emergency department units and emergency medical services
* Age ≥ 18 years

Exclusion Criteria:

* Inability to participate in all aspects of the study prior to study begin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Tests of Knowledge of the FAST Examination | 1 day
  knowledge-based measures used to evaluate participants' knowledge of FAST-examination-related concepts (Survey)

SECONDARY OUTCOMES:
FAST Performance Test | 1 day
  The performance test required participants to conduct a FAST examination on two model patients (one normal, one ascites positive). No help or feedback was given to the participants.
Window acquisition time | 1 day
  Identification of FAST Window Quadrants and Diagnostic Interpretation of FAST Windows.
  The window acquisition time was measured with a stopwatch and represented the period between first contact of the probe with the model patient's body and when the participant said "stop" to indicate an adequate window or the participant's judgment that he or she could not acquire the window.
Window quality | 1 day
  For each acquired window, an expert evaluated the quality of the window. The window was rated as "excellent, fair, poor, or other." "Other" captured situations where the window acquired was nondiagnostic. Window quality was dichotomized into two categories, "excellent or not excellent," and subsequent analyses examined the number of participants that acquired "excellent" windows by quadrant (perihepatic space (also called Morison's pouch or the hepatorenal recess), perisplenic space, pericardium, and the pelvis and suprapubic quadrant) and patient type (normal, positive).
Diagnostic accuracy | 1 day
  For each acquired window, the participant rendered a diagnosis of that window. An expert evaluated the quality of the diagnosis. The diagnosis was rated as "correct, incorrect, or other." "Other" captured situations where the window acquired was nondiagnostic. For analysis purposes, diagnostic accuracy was dichotomized into two categories, "correct or not correct," and subsequent analyses examined the number of participants that interpreted the window correctly by quadrant (perihepatic space (also called Morison's pouch or the hepatorenal recess), perisplenic space, pericardium, and the pelvis and suprapubic quadrant) and patient type (normal, positive).

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Principal Investigator — Institute of Cardiology
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Poland